CLINICAL TRIAL: NCT02904954
Title: A Randomized Phase 2 Trial of Durvalumab (MEDI4736) With or Without SBRT in Clinical Stage I, II, and IIIA Non-small Cell Lung Cancer (NSCLC)
Brief Title: Durvalumab (MEDI4736) With or Without SBRT in Clinical Stage I, II and IIIA Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1501015795
Record Dates: First submitted 2016-05-18; First posted 2016-09-19 (Estimated); Results first posted 2021-08-03 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-01

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Lung neoplasms; Bronchial Neoplasms; Carcinoma, bronchogenic; Neoplasms; Neoplasms by site; Respiratory Tract Diseases; Respiratory Tract Neoplasms; Thoracic Neoplasms
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Bronchial Neoplasms; Carcinoma, Bronchogenic; Neoplasms; Neoplasms by Site; Respiratory Tract Diseases; Respiratory Tract Neoplasms; Thoracic Neoplasms | interventions — durvalumab; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Durvalumab monotherapy) (Experimental): Durvalumab (MEDI4736) 1.12 g administered pre-operatively every 3 weeks for 2 cycles followed by surgical resection. Durvalumab monotherapy 1.5 g will be given for 12 months post-operatively.
  Interventions: Drug: Durvalumab
- Arm 2 (Durvalumab plus SBRT) (Experimental): Durvalumab (MEDI4736) 1.12 g administered pre-operatively every 3 weeks for 2 cycles plus radiotherapy delivered in 3 daily fractions starting concurrently with the first cycle of durvalumab (MEDI4736) followed by surgical resection. Durvalumab monotherapy 1.5 g will be given for 12 months post-operatively.
  Interventions: Drug: Durvalumab; Other: Durvalumab plus SBRT

INTERVENTIONS:
Drug: Durvalumab — Intravenously
  Other Names: MEDI4736
Other: Durvalumab plus SBRT — Intravenously plus radiotherapy
  Other Names: MEDI4736
  Arms: Arm 2 (Durvalumab plus SBRT)

SUMMARY:
The purpose of this study is to find out the effectiveness of the drug durvalumab (MEDI4736) with or without stereotactic body radiation therapy (SBRT) as treatment for stage I (tumors > 2cm), II, and IIIA non-small cell lung cancer (NSCLC) prior to surgery and one year following surgery.

DETAILED DESCRIPTION:
This is a randomized open label phase II trial of preoperative anti-PD-L1 antibody durvalumab with or without concurrent non-ablative radiation followed by surgical resection and postoperative monthly maintenance durvalumab for twelve months, following standard of care postoperative therapy.

ELIGIBILITY:
Inclusion Criteria

1. Patient has histologically or cytologically proven clinical stages I (tumors > 2 cm), II, and IIIA NSCLC and is considered eligible for surgical resection with curative intent. Patients with 2 primary non-small cell lung cancers are allowed.
2. Measureable disease, as defined by RECIST v1.1.
3. Written informed consent and HIPAA obtained from the subject prior to performing any protocol-related procedures.
4. Age > 18 years at time of study entry
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
6. Adequate normal organ and marrow function as defined below:

   * Haemoglobin ≥ 9.0 g/dL
   * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L (> 1500 per mm3)
   * Platelet count ≥ 100 x 109/L (>100,000 per mm3)
   * Serum bilirubin ≤ 1.5 x institutional upper limit of normal (ULN). This will not apply to subjects with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only in consultation with their physician.
   * AST (SGOT)/ALT (SGPT), and alkaline phosphatase ≤ 2.5 x institutional upper limit of normal (ULN).
   * Serum creatinine CL>40 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance:
7. Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal patients. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

   Women <50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy).

   Women ≥50 years of age would be considered post-menopausal if they have been amenorrheic exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, had chemotherapy-induced menopause with last menses >1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).
8. Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
9. No prior therapy for their lung cancer.

Exclusion Criteria

Subjects should not enter the study if any of the following exclusion criteria are fulfilled:

1. Participation in another clinical study with an investigational product during the last 3 weeks.
2. History of another primary malignancy except for:

   * Malignancy treated with curative intent and with no known active disease ≥3 years before the first dose of study drug and of low potential risk for recurrence.
   * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease.
   * Adequately treated carcinoma in situ without evidence of disease eg, cervical cancer in situ, in-situ urinary bladder cancer , treated localized prostate cancer and ductal carcinoma-in situ.
   * Indolent hematological malignancies
3. Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab, with the exceptions of intranasal,inhaled, topical steroids, or local steroid injections (e.g., intra articular injection), corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid, and steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication).
4. Any unresolved toxicity (CTCAE grade 2) from therapy for a prior malignancy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria.

   * Patients with Grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the Study Physician.
   * Subjects with irreversible toxicity that is not reasonably expected to be exacerbated by the investigational product may be included (e.g., hearing loss, peripherally neuropathy).
5. Any prior Grade ≥3 immune-related adverse event (irAE) while receiving any previous immunotherapy agent, or any unresolved irAE >Grade 1.
6. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). No active diverticulitis within the previous 3 months. The following are exceptions to this criterion:

   * Patients with vitiligo or alopecia
   * Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
   * Any chronic skin condition that does not require systemic therapy
   * Patients without active disease in the last 5 years may be included but only after consultation with the study physician
   * Patients with celiac disease controlled by diet alone
7. Active or prior documented inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis).
8. History of active primary immunodeficiency.
9. History of allogeneic organ transplant.
10. History of hypersensitivity to durvalumab or any excipient.
11. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent.
12. Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), hepatitis B (known positive HBV surface antigen (HBsAg) result), hepatitis C, or human immunodeficiency virus (positive HIV 1/2 antibodies). Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
13. History of leptomeningeal carcinomatosis.
14. Receipt of live attenuated vaccination within 30 days prior to study entry or within 30 days of receiving durvalumab.
15. Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of durvalumab monotherapy.
16. Any condition that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study results
17. Subjects with uncontrolled seizures.
18. History of interstitial lung disease, idiopathic pulmonary fibrosis, pneumonitis (including drug induced), or evidence of active pneumonitis on screening chest CT scan.
19. Major surgical procedure within 28 days prior to Cycle 1, Day 1 or anticipation of need for a major surgical procedure during the course of the study.
20. Receipt of the last dose of therapy (chemotherapy, immunotherapy, endocrine therapy, targeted therapy, biologic therapy, tumor embolization, monoclonal antibodies, or other investigational agent) for an accepted other malignancy as defined in Section 3.3.2 within 30 first dose of study drug for lung cancer.
21. Prior randomisation or treatment in a previous durvalumab clinical study regardless of treatment arm assignment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-12-02 (Actual); Primary Completion 2020-09-16 (Actual); Study Completion 2022-10-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nasser K Altorki, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Altorki NK, Walsh ZH, Melms JC, Port JL, Lee BE, Nasar A, Spinelli C, Caprio L, Rogava M, Ho P, Christos PJ, Saxena A, Elemento O, Bhinder B, Ager C, Amin AD, Sanfilippo NJ, Mittal V, Borczuk AC, Formenti SC, Izar B, McGraw TE. Neoadjuvant durvalumab plus radiation versus durvalumab alone in stages I-III non-small cell lung cancer: survival outcomes and molecular correlates of a randomized phase II trial. Nat Commun. 2023 Dec 19;14(1):8435. doi: 10.1038/s41467-023-44195-x. PMID 38114518
- [Derived] Lee B, Mynard N, Nasar A, Villena-Vargas J, Chow O, Harrison S, Stiles B, Port J, Altorki N. Surgical resection after neoadjuvant durvalumab and radiation is feasible and safe in non-small cell lung cancer: Results from a randomized trial. J Thorac Cardiovasc Surg. 2023 Jan;165(1):327-334.e2. doi: 10.1016/j.jtcvs.2022.07.017. Epub 2022 Aug 6. PMID 36028357
- [Derived] Altorki NK, McGraw TE, Borczuk AC, Saxena A, Port JL, Stiles BM, Lee BE, Sanfilippo NJ, Scheff RJ, Pua BB, Gruden JF, Christos PJ, Spinelli C, Gakuria J, Uppal M, Binder B, Elemento O, Ballman KV, Formenti SC. Neoadjuvant durvalumab with or without stereotactic body radiotherapy in patients with early-stage non-small-cell lung cancer: a single-centre, randomised phase 2 trial. Lancet Oncol. 2021 Jun;22(6):824-835. doi: 10.1016/S1470-2045(21)00149-2. Epub 2021 May 18. PMID 34015311

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 64 enrolled participants, 60 met inclusion criteria and were randomized to treatment.
Groups:
- Arm 2 (Durvalumab Plus SBRT): Durvalumab (MEDI4736) 1.12 g administered pre-operatively every 3 weeks for 2 cycles plus radiotherapy delivered in 3 daily fractions starting concurrently with the first cycle of durvalumab (MEDI4736) followed by surgical resection. Durvalumab monotherapy 1.5 g will be given for 12 months post-operatively.
  Durvalumab: Intravenously
  Durvalumab plus SBRT: Intravenously
Period: Neoadjuvant (Preoperative) to Surgery
Arm/Group | Arm 1 (Durvalumab Monotherapy) | Arm 2 (Durvalumab Plus SBRT)
Started | 30 | 30
Completed | 26 (30 participants completed 2 neoadjuvant cycles. Surgical resection was not performed in 4 participants.) | 26 (30 participants completed the first neoadjuvant Durvalumab cycle combined with SBRT. Three subjects did not receive the 2nd cycle. Surgical resection was not performed in 4 participants.)
Not Completed | 4 | 4
Not completed — Death | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Disease progression | 2 | 3
Period: Adjuvant Durvalumab
Arm/Group | Arm 1 (Durvalumab Monotherapy) | Arm 2 (Durvalumab Plus SBRT)
Started | 26 | 26
Completed | 6 | 11
Not Completed | 20 | 15
Not completed — Recurrence | 2 | 0
Not completed — Adverse Event | 2 | 6
Not completed — Participant wishes | 12 | 7
Not completed — Physician Decision | 2 | 1
Not completed — Slow recovery after chemotherapy | 1 | 0
Not completed — Death | 0 | 1
Not completed — Prostate cancer | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm 1 (Durvalumab Monotherapy): Durvalumab (MEDI4736) via IV infusion administered pre-operatively every 3 weeks for 2 cycles followed by surgical resection. Durvalumab monotherapy will be given for 12 months post-operatively.
  Durvalumab: Intravenously
- Arm 2 (Durvalumab Plus SBRT): Durvalumab (MEDI4736) via IV infusion administered pre-operatively every 3 weeks for 2 cycles plus radiotherapy delivered in 3 daily fractions starting concurrently with the first cycle of durvalumab (MEDI4736) followed by surgical resection. Durvalumab monotherapy will be given for 12 months post-operatively.
  Durvalumab: Intravenously
  Durvalumab plus SBRT: Intravenously
- Total: Total of all reporting groups
Arm/Group | Arm 1 (Durvalumab Monotherapy) | Arm 2 (Durvalumab Plus SBRT) | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.5 (7.5) | 69.6 (9.4) | 70.2 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 15 | 29
  Male | 16 | 15 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 6 | 6
  Not Hispanic or Latino | 30 | 24 | 54
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 4 | 7
  White | 25 | 23 | 48
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Major Pathological Response (MPR)
Description: MPR is defined as ≤10% residual viable tumor in the resected specimen.
Time Frame: Durvalumab start date to surgical resection, up to 10 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 (Durvalumab Monotherapy) | Arm 2 (Durvalumab Plus SBRT)
Number analyzed (Participants) | 30 | 30
Participants | 2 | 16
Statistical Analysis 1: Comparison: Arm 1 (Durvalumab Monotherapy) vs Arm 2 (Durvalumab Plus SBRT); Fisher's exact test performed to compare the MPR proportion between the two treatment arms. Null hypothesis is that there is no difference in the MPR proportion between the two arms; Test type: Superiority; p = 0.0001, Fisher Exact — Testing at alpha = 0.05; Risk Difference (RD) = 46.6, 95% CI 2-sided [26.7 to 66.6]

2. Secondary Outcome: Kaplan-Meier Disease-Free Survival Proportion at 2 Years
Description: Disease recurrence or death from any cause assessed using history, physical examination and CT scanning, histologically or cytologically confirmed whenever possible.
Time Frame: From date of Durvalumab start date until the date of first documented progression or date of death from any cause, whichever came first, assessed every 6 months for 2 years.
Measure: Number (95% Confidence Interval); unit: Proportion of subjects
Arm/Group | Arm 1 (Durvalumab Monotherapy) | Arm 2 (Durvalumab Plus SBRT)
Number analyzed (Participants) | 30 | 30
Proportion of subjects | 0.67 [0.50 to 0.84] | 0.80 [0.66 to 0.94]
Statistical Analysis 1: Comparison: Arm 1 (Durvalumab Monotherapy) vs Arm 2 (Durvalumab Plus SBRT); Kaplan-Meier survival analysis comparing the two arms; Test type: Superiority; p = 0.89, Log Rank

3. Secondary Outcome: Objective Clinical Response Rate
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by PET/CT scan: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of diameters of target lesions; Progressive Disease (PD), >=20% increase in the sum of diameters of target lesions; Stable Disease (SD), neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD.
Time Frame: Treatment day 1 up to weeks 6-7
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 (Durvalumab Monotherapy) | Arm 2 (Durvalumab Plus SBRT)
Number analyzed (Participants) | 30 | 30
Participants
  Complete Response | 0 | 0
  Partial Response | 1 | 14
  Progressive Disease | 3 | 1
  Pseudoprogression | 2 | 0
  Stable Disease | 24 | 15
Statistical Analysis 1: Comparison: Arm 1 (Durvalumab Monotherapy) vs Arm 2 (Durvalumab Plus SBRT); Fisher's exact test performed to compare the objective clinical response proportion between the two treatment arms. Null hypothesis is that there is no difference in the objective clinical response proportion between the two arms. Objective clinical response proportion is defined as the proportion of patients in each arm who have complete response or partial response; Test type: Superiority; p = 0.0001, Fisher Exact — Testing at alpha = 0.05; Risk Difference (RD) = 43.4, 95% CI 2-sided [24.4 to 62.3]

4. Other Pre Specified Outcome: Number of Participants With Treatment-related Adverse Events as Assessed by CTCAE v. 4.0
Description: Adverse events ≥G3 in both arms with and without possible or probable attribution to study drug and graded according to CTCAE v. 4.0
Time Frame: Up to 72 weeks
Population: All randomized patients
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 (Durvalumab Monotherapy) | Arm 2 (Durvalumab Plus SBRT)
Number analyzed (Participants) | 30 | 30
Participants | 12 | 15

ADVERSE EVENTS:
Time Frame: From enrollment to 90 days after the last dose of durvalumab
Arm/Group | Arm 1 (Durvalumab Monotherapy) | Arm 2 (Durvalumab Plus SBRT)
All-Cause Mortality (participants affected / at risk) | 9/30 | 10/30
Serious Adverse Events (participants affected / at risk) | 12/30 | 15/30
Other Adverse Events (participants affected / at risk) | 29/30 | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (Durvalumab Monotherapy) (N=30) | Arm 2 (Durvalumab Plus SBRT) (N=30)
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 1 | 0
Stroke (Nervous system disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Cardiopulmonary event (Cardiac disorders) | 0 | 1
Thromboembolic event (Vascular disorders) | 3 | 5
Platelet count decreased (Investigations) | 0 | 1
Hyponatremia (Investigations) | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Anaphylaxis (Immune system disorders) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 0 | 2
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Atrial flutter (Cardiac disorders) | 1 (1) | 0
Autoimmune hemolytic anemia (Immune system disorders) | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 1
Bronchopleural Fistula (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Fatigue (General disorders) | 1 | 3
Heparin induced thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Lung infection (Infections and infestations) | 1 | 8
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Seroma (Injury, poisoning and procedural complications) | 0 | 1
Surgical wound infection (Infections and infestations) | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pericarditis (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 2
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 (Durvalumab Monotherapy) (N=30) | Arm 2 (Durvalumab Plus SBRT) (N=30)
Constipation (Gastrointestinal disorders) | 20 | 21
Fatigue (General disorders) | 18 | 14
Anemia (Blood and lymphatic system disorders) | 10 | 16
Cough (Respiratory, thoracic and mediastinal disorders) | 13 | 13
Nausea (Gastrointestinal disorders) | 9 | 11
Diarrhea (Gastrointestinal disorders) | 10 | 9
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8 | 12
Hypotension (Vascular disorders) | 8 | 9
Lipase increased (Investigations) | 8 | 10
Serum amylase increased (Investigations) | 6 | 8
Anorexia (Metabolism and nutrition disorders) | 4 | 7
Rash (Skin and subcutaneous tissue disorders) | 5 | 6
Hyperkalemia (Investigations) | 5 | 5
Urinary tract infection (Infections and infestations) | 3 | 5
Hyperglycemia (Investigations) | 2 | 7
Fever (General disorders) | 3 | 4
Hypertension (Vascular disorders) | 3 | 3
Vomiting (Gastrointestinal disorders) | 3 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 6
Pruritis (Skin and subcutaneous tissue disorders) | 1 | 6
Hypoalbuminemia (Investigations) | 2 | 5
Dizziness (Nervous system disorders) | 2 | 4
Headache (Nervous system disorders) | 3 | 5
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 3
Alkaline phosphatase increased (Investigations) | 1 | 4
Atrial fibrillation (Cardiac disorders) | 2 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 2
Chills (General disorders) | 1 | 4
Infusion related reaction (General disorders) | 2 | 3
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Aspartate aminotransferase increased (Investigations) | 1 | 3
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 2
Hyperthyroidism (Endocrine disorders) | 3 | 1
Hypothyroidism (Endocrine disorders) | 4 | 0
Presyncope (Nervous system disorders) | 2 | 2
Weight loss (Investigations) | 2 | 2
Hyponatremia (Investigations) | 3 | 0
Alanine aminotransferase increased (Investigations) | 2 | 1
Platelet count decreased (Investigations) | 2 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 3
Colitis (Gastrointestinal disorders) | 2 | 0
Immune related thyroiditis (Endocrine disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-03): https://cdn.clinicaltrials.gov/large-docs/54/NCT02904954/Prot_SAP_002.pdf